CLINICAL TRIAL: NCT05788627
Title: Effectiveness Of Oral Lactulose Versus Lactulose Enema On The Time To Recovery From Overt Hepatic Encephalopathy
Brief Title: Effectiveness of Oral Lactulose Versus Lactulose Enema in Hepatic Encephalopathy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Khyber Medical College, Peshawar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 700
Record Dates: First submitted 2023-03-14; First posted 2023-03-29 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Hepatic Encephalopathy; Chronic Liver Disease
MeSH Terms: conditions — Hepatic Encephalopathy | interventions — Lactulose

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo arm / tap water enema arm (Placebo Comparator): This arm will receive oral lactulose as per treatment protocol for hepatic encephalopathy i.e. 30ml twice daily. And will receive tap water enema as placebo i.e. 1000ml tap water enema twice daily.
  Interventions: Drug: Tap water
- Lactulose enema arm (Experimental): This arm will receive oral lactulose in a dose of 30ml twice daily alongwith lactulose enema (300ml lactulose plus 700ml water) twice daily.
  Interventions: Drug: Lactulose

INTERVENTIONS:
Drug: Tap water — Oral lactulose in a dose of 30ml BD and tap water enema 1000ml BD
  Other Names: tap water enema
  Arms: Placebo arm / tap water enema arm
Drug: Lactulose — Oral lactulose in a dose of 30ml BD and lactulose enema (300ml lactulose and 700ml water) in a dose of 1000ml BD.
  Other Names: Lactulose enema
  Arms: Lactulose enema arm

SUMMARY:
Patients with chronic liver disease due to hepatitis B or C viruses, Non-alcoholic fatty liver disease, autoimmune hepatitis, wilson disease, cryptogenic hepatitis etc are prone to develop complications. Hepatic encephalopathy is one of such complications. It is graded into four types depending on severity of clinical features, which range through altered sleep pattern to coma. The current study aims to compare the effectiveness of lactulose enema with oral lactulose in time to recovery from higher grade of encephalopathy to lower grade of encephalopathy.

DETAILED DESCRIPTION:
Hepatic encephalopathy (HE) is defined as neuropsychiatric disorder due to liver failure. It is characterized by mild cognitive impairment, stupor and coma. The most common reasons for pathogenesis include the role of neurotoxins, impaired neurotransmission due to metabolic changes in liver failure, changes in brain energy metabolism, systemic inflammatory response and alterations of the blood brain barrier. Neurotoxin ammonia is related to precipitating HE, for which the gastrointestinal tract is the primary source. Colonic bacteria catabolise the nitrogenous sources into ammonia.

Lactulose is the initial treatment for HE. It produces diarrhea by osmosis and reduces pH of colonic contents, which leads to reduced absorption of ammonia by converting it to ammonium ion (NH4). Understandingly, it does not cure the underlying liver disease however, it does prevent deterioration of the mental status in HE.

Initial oral dose of lactulose is 30 ml once a day or twice daily. For retention enema the dose is 300 ml lactulose plus 700 ml water, administered every 4 hours. It can be increased as tolerated. At least, 2-4 loose stools per day should be passed by the patient.

Lactulose is also effective as primary prophylaxis against the development of HE.

Constipation is one very common precipitating factor for hepatic encephalopathy which is routinely managed with oral lactulose or kleen enema (21.4g (18.1% w/v) Sodium Dihydrogen Phosphate Dihydrate and 9.4g (8.0% w/v) Disodium Phosphate Dodecahydrate). Lactulose enema is also given to patients in hepatic encephalopathy either alone or in combination with oral lactulose. However it is not clear whether there is any difference in the efficacy of oral or enema lactulose in patients with hepatic encephalopathy in terms of improvement of encephalopathy grade and time to improvement. This study aims to determine the efficacy of oral versus enema lactulose in the achievement of these goals.

ELIGIBILITY:
Inclusion Criteria:

* Male and female cirrhotic patients in grades 3 or 4 of hepatic encephalopathy
* Patient with constipation as the precipitating factor will be included in the study

Exclusion Criteria:

* Patients with dehydration
* Electrolyte abnormalities
* Spontaneous bacterial peritonitis (SBP),
* Fever
* Using sedative / hypnotic medications as predisposing factors for hepatic encephalopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Change in grade of hepatic encephalopathy | Over 48 hours
  Change in HE grade from grade 4 to grade 3 or grade 3 to grade 2

SECONDARY OUTCOMES:
Relief of constipation | Over 48 hours
  Frequency of 2-3 soft stools per 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Aliena Badshah, Principal Investigator — Khyber Medical College

IPD SHARING:
Plan to Share IPD: Yes
Patients confidentiality shall be maintained at all stages. Other patient characteristics e.g grade of encephalopathy, serum ammonia levels before and after initiation of intervention, response to lactulose enema can be shared if required.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will become available once patients are recruited into the study
Access Criteria: not specified yet